CLINICAL TRIAL: NCT00000307
Title: Naltrexone as an Adjunct in Alcoholic Cocaine Dependent Patients
Brief Title: Naltrexone as Adjunct in Alcoholic Cocaine Dependent Patients - 4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Texas (Other)
Responsible Party: Joy Schmitz, Ph.D., University of Texas Medical School at Houston
Purpose: Treatment
Other Study IDs: NIDA-09262-4; P50-09262-4
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol-Related Disorders; Cocaine-Related Disorders
Keywords: alcohol dependence
MeSH Terms: conditions — Alcohol-Related Disorders; Cocaine-Related Disorders; Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Naltrexone

SUMMARY:
The purpose of this study is to evaluate naltrexone as an adjunct in alcoholic cocaine dependent patients; concurrent relapse prevention theory.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 2003-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Verified abstinence from cocaine | over the 12 weeks of study

CONTACTS AND LOCATIONS:
Overall Officials: John Grabowski, Ph.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States